CLINICAL TRIAL: NCT01817465
Title: A Multi-centers, Randomized, Double-blinded, Parallel Study Study to Evaluate the Efficacy and Safety of Motilitone® in Patients With Functional Dyspepsia.
Brief Title: A Study to Demonstrate the Efficacy and Safety of Motilitone®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DA9701_PPI_IV
Record Dates: First submitted 2013-03-19; First posted 2013-03-25 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Motilione® (Experimental): 30 mg is administered with a tablet of placebo (Pantoline®)
  Interventions: Drug: Motilitone ®
- Pantoline® (Active Comparator): 40mg is administered with a tablet of Motilitone®
  Interventions: Drug: Pantoline®
- Motilitone® and Pantoline® (Active Comparator): Both drugs are administered at once
  Interventions: Drug: Motilitone® and Pantoline®

INTERVENTIONS:
Drug: Motilitone ®
  Arms: Motilione®
Drug: Pantoline®
  Arms: Pantoline®
Drug: Motilitone® and Pantoline®
  Arms: Motilitone® and Pantoline®

SUMMARY:
This is a phase IV , comparative study to evaluate the efficacy and safety of Motiltone® in treatment of the patients with functional dyspepsia. The study is conducted with following methods: multi-centers, double blind, randomization, parallel. The subjects will receive Motilitone® or/and Pantoline®.

ELIGIBILITY:
Inclusion Criteria:

* Roman III criteria
* One or more conditions are applied: epigastralgia, burning feelings in the solar plexus early satiety, uncomfortable fullness
* No organic lesion

Exclusion Criteria:

* has been administered or was administered within a month
* had a surgery that might affect gastrointestinal motility
* Tegaserod

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2012-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Subject global assessment by using 5-Likert scale and Binary outcome methods | 6 weeks
  5-Likert scale: 0: worse
  1. similar
  2. improved in some degree
  3. considerably improved
  4. completely cured
  Binary outcome:
  yes/no

SECONDARY OUTCOMES:
Number of dyspepsia(indigestion) symptoms occurred (Counted daily) | 6 weeks
Assessment of NDI-K Quality of Life | 6 weeks
Soreness of digestive symptoms (dyspepsia) evaluated its intensity on a scale of 1 to 5 | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Myung Kyu Choi, M.D., Ph.D., Principal Investigator — The Catholic University of Korea; Kyu Chan Huh, M.D., Ph.D., Principal Investigator — Konyang University Hospital; Sung Kook Kim, M.D., Ph.D., Principal Investigator — Kyungpook National University Hospital; Kyung Sik Park, M.D., Ph.D., Principal Investigator — Keimyung University Dongsan Medical Center; Joong Gu Gweon, M.D.,Ph.D., Principal Investigator — Daegu Catholic University Medical Center; Geun Am Song, M.D., Ph.D., Principal Investigator — Busan National University Hospital; Soo Jin Hong, M.D., Ph.D., Principal Investigator — Soonchunhyang University Hospital; Na Young Kim, M.D., Ph.D., Principal Investigator — Seoul National University Bundang Hospital; Jung Il Son, M.D., Ph.D., Principal Investigator — Kangbuk Samsung Hospital; Poong Yul Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center; Joon Sung Lee, M.D., Ph.D., Principal Investigator — Soonchunhyang University Hospital; Hoon Yong Jung, M.D., Ph.D., Principal Investigator — Asan Medical Center; Hyo Jin Park, M.D., Ph.D., Principal Investigator — Gangnam Severance Hospital; Yong Chan Lee, M.D., Ph.D., Principal Investigator — Severance Hospital; Suk Chae Choi, M.D., Ph.D., Principal Investigator — Wonkwang Medical Center; Hye Kyung Jung, M.D., Ph.D., Principal Investigator — Iwha Womans Unversity Mokdong Hospital; Sam Ryong Ji, M.D., Ph.D., Principal Investigator — Inje University; Jong Sun Ryu, M.D., Ph.D., Principal Investigator — Chonnam National University Hospital; Oh Young Lee, M.D., Ph.D., Principal Investigator — Hanyang University
Locations (1):
- Ajou University Medical Center, Suwon, South Korea